CLINICAL TRIAL: NCT03068312
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Efficacy of Ivacaftor in Subjects With Cystic Fibrosis Who Are 6 Years of Age and Older and Have Either a 3849 + 10KB C→T or D1152H-CFTR Mutation
Brief Title: A Study to Evaluate Efficacy of Ivacaftor in Subjects With Cystic Fibrosis Who Have a 3849 + 10KB C→T or D1152H CFTR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX16-770-127; 2017-000457-39 (EudraCT Number)
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Results first posted 2020-01-06 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sequence 1: First Ivacaftor (IVA) Then Placebo (Experimental): Participants received IVA 150 milligram (mg) every 12 hours (q12h) for 8 weeks in treatment period 1 followed by placebo matched to IVA for 8 weeks in treatment period 2. A washout period of 8 weeks was maintained between the 2 treatment periods.
  Interventions: Drug: Ivacaftor; Drug: Placebo
- Sequence 2: First Placebo Then IVA (Experimental): Participants received placebo matched to IVA for 8 weeks in treatment period 1 followed by IVA 150 mg q12h for 8 weeks in treatment period 2. A washout period of 8 weeks was maintained between the 2 treatment periods.
  Interventions: Drug: Ivacaftor; Drug: Placebo

INTERVENTIONS:
Drug: Ivacaftor — IVA 150 mg tablet.
  Other Names: VX-770; IVA
Drug: Placebo — Placebo matched to IVA tablet.

SUMMARY:
This study will evaluate the efficacy of ivacaftor treatment in subjects with CF 6 years of age and older who have a 3849 + 10KB C→T or D1152H CFTR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF based on protocol-specified clinical features and at least one of the following: increased sweat chloride level, identification of 2 CF causing mutations, or demonstration of abnormal nasal epithelial ion transport.
* A 3849 + 10KB C→T or D1152H mutation on at least 1 CFTR allele.
* FEV1 ≥40% of predicted and ≤105% of predicted at screening.

Exclusion Criteria:

* A G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549N, S549R, or R117H mutation.
* History of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Ongoing or prior participation in an investigational drug study within 30 days before the Screening Visit.
* Protocol-specified abnormal laboratory values at the Screening Visit
* For subjects <18 years of age at the Screening Visit, evidence of cataract/lens opacity determined to be clinically significant by the ophthalmologist or optometrist during the ophthalmologic examination (OE) at the Screening Visit.
* Use of any moderate or strong inducers or inhibitors of cytochrome P450 (CYP) 3A, including consumption of certain herbal medications and certain fruit and fruit juices, within 14 days before Day 1.
* Pregnant, breastfeeding, or planning to become pregnant during the study.
* Sexually active subjects of reproductive potential must be willing to use appropriate contraception.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Kerem E, Cohen-Cymberknoh M, Tsabari R, Wilschanski M, Reiter J, Shoseyov D, Gileles-Hillel A, Pugatsch T, Davies JC, Short C, Saunders C, DeSouza C, Sullivan JC, Doyle JR, Chandarana K, Kinnman N. Ivacaftor in People with Cystic Fibrosis and a 3849+10kb C-->T or D1152H Residual Function Mutation. Ann Am Thorac Soc. 2021 Mar;18(3):433-441. doi: 10.1513/AnnalsATS.202006-659OC. PMID 33095038

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF).
Period: Overall Study
Arm/Group | Sequence 1: First Ivacaftor (IVA) Then Placebo | Sequence 2: First Placebo Then IVA
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: First IVA Then Placebo: Participants received IVA 150 mg q12h for 8 weeks in treatment period 1 followed by placebo matched to IVA for 8 weeks in treatment period 2. A washout period of 8 weeks was maintained between the 2 treatment periods.
- Total: Total of all reporting groups
Arm/Group | Sequence 1: First IVA Then Placebo | Sequence 2: First Placebo Then IVA | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (15.3) | 32.1 (15.6) | 32.3 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Lung Clearance Index 2.5 (LCI2.5) [Mean (Standard Deviation); unit: lung clearance index] — LCI2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
  lung clearance index | 12.74 (4.04) | 13.19 (5.45) | 12.96 (4.74)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lung Clearance Index 2.5 (LCI2.5)
Description: LCI2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
Time Frame: From baseline through 8 weeks
Population: The Full Analysis Set (FAS) included all randomized subjects who carried the intended CFTR allele mutation and received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: lung clearance index
Groups:
- Placebo: All participants who received placebo matched to IVA for 8 weeks in treatment period 1 or 2.
- Ivacaftor: All participants who received IVA for 8 weeks in treatment period 1 or 2.
Arm/Group | Placebo | Ivacaftor
Number analyzed (Participants) | 37 | 37
lung clearance index | 0.20 (0.19) | -0.46 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Ivacaftor; Test type: Other; Least squares mean difference = -0.66, 95% CI 2-sided [-1.10 to -0.21]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to safety follow-up visit (up to Week 28)
Arm/Group | Placebo | Ivacaftor
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 2/38 | 1/38
Other Adverse Events (participants affected / at risk) | 19/38 | 12/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | Ivacaftor (N=38)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | Ivacaftor (N=38)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Headache (Nervous system disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 2
Malaise (General disorders) | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 2 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Viral upper respiratory tract infection (Infections and infestations) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT03068312/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT03068312/SAP_001.pdf